CLINICAL TRIAL: NCT01819558
Title: Etude Phase I/II d'immunothérapie Par protéine recWT1-A10+AS01B après Greffe allogénique de Cellules Souches
Brief Title: Phase I/II Study of Immune Therapy After Allograft in Patients With Myeloid Hemopathy
Acronym: ALLO-WT1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-WT1/IPC 2011-006
Record Dates: First submitted 2013-03-19; First posted 2013-03-27 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: acute myeloid leukemia; chronic myeloid leukemia; myelodysplastic syndrome; allograft; WT1 expression
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes | interventions — Immunotherapy, Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- immune therapy (Experimental): 6 administration every 2 weeks of intra-muscular 200 micrograms of protein recwt1-A10+AS01B at week 1, 3, 5, 7, 9 and 11.
  Interventions: Biological: recwt1-A10+AS01B

INTERVENTIONS:
Biological: recwt1-A10+AS01B
  Other Names: immune therapy

SUMMARY:
Patients with acute or chronic myeloid leukemia, or myelodysplastic syndrome, underwent allogeneic stem cell transplantation from HLA-identical donor (related or unrelated) after reduced-intensity conditioning regimen.

If WT1 expression is detectable on tumor cells, they will receive an immune therapy 60 days after allograft.

6 administrations every 2 weeks of the protein recwt1-A10+AS01B will be administrated.

The safety and immunological efficacy of this immune therapy after hematopoietic stem cells transplantation with reduced intensity conditioning will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 and younger than 65 years.
2. Karnofsky ≥ 70 %.
3. Patients with acute or chronic myeloid leukemia, or myelodysplastic syndrome, who underwent allogeneic stem cell transplantation from HLA-identical donor (related or unrelated) after reduced-intensity conditioning regimen.
4. Patients in morphologic complete remission at the time of transplantation.
5. WT1 expression detectable on tumor cells.
6. Expected life duration more than 6 months.
7. Creatinine clearance ≥ 50 ml/min
8. Bilirubinemia < 1.5N and ASAT < 2.5N.
9. Women of childbearing age: negative pregnancy test and effective contraception for at least 30 days before vaccinal immunotherapy (the same contraceptive method must be continued at least 2 months after the last vaccine infusion).
10. Membership of a social security scheme or beneficiary of such a regime.
11. Signed inform consent.

Exclusion Criteria:

1. Patients with severe and uncontrolled affections, especially active graft-versus-host disease requiring steroid treatment (>0.3 mg/kg/j) and/or Mycophenolate mofetil.
2. Pregnant or lactating women.
3. HIV seropositive patients.
4. Autoimmune disease (Lupus, multiple sclerosis, Chron disease…)
5. Previous history of allergic state which could be potentially compound by a component of the vaccinal immunotherapy.
6. Patients who received (or are planned to receive) another experimental treatment within 30 days following the first infusion of the experimental drug of this protocol.
7. Previous history of another cancer, except if considered as probably cured by the investigator.
8. Patients deprived of liberty, or under guardianship.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
safety | 30 days
  Dose limit toxicity (adverse event according to CTCAE V4.0)

SECONDARY OUTCOMES:
immune response | up to 60 weeks after treatment
  The specific WT1 antibody induced by the vaccination will be evaluated by the technic ELISA in UE/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Didier BLAISE, MD PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr/